CLINICAL TRIAL: NCT06218992
Title: Corneal and Tear Film Changes in Chinese Patients With Type 2 Diabetes: a Cross-sectional Controlled Study
Brief Title: Corneal and Tear Film Changes in Chinese Patients With Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DM2023
Record Dates: First submitted 2024-01-10; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease; Tear Film; Corneal Nerve
Keywords: dry eye; tear film
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Type 2 diabetic patients
- Control group: Age- and sex-matched subjects without DM

SUMMARY:
Diabetes mellitus has been associated with ocular surface damage and exacerbates dry eye disease (DED) pathology. To investigate clinical and inflammatory changes in the ocular surface of insulin-independent type II diabetic patients. This cross-sectional control study will recruit 200 Type 2 diabetic patients and 200 age- and sex-matched subjects without DM.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a developing global health challenge due to the multiple complications associated with long-term hyperglycemia. Although diabetic retinopathy is the most prevalent and well-known ophthalmic consequence, diabetes also causes clinically significant effects on the ocular surface. Among the ocular surface diseases, dry eye disease (DED) is the most common. Multiple mechanisms, such as ocular surface and lacrimal gland inflammation, neurotrophic deficiency, and meibomian gland dysfunction (MGD), play significant roles.

A loss of tear film homeostasis characterizes DED. DM is one of the risk factors for DED; 47% of DM patients suffer from ocular surface damage due to negative alterations to the tear film, corneal thickness, corneal epithelium, corneal nerve, and corneal endothelium. It has been suggested that one or more of the following initial events may lead to alterations described in the tear film and ocular surface of patients with DM: a) chronic hyperglycemia, b) corneal nerve damage, and c) impairment on insulin action.

Previous studies have explored the association between DM and ocular surface dysfunction. However, ocular surface and tear film parameters in diabetic patients are lacking in the Chinese population. Moreover, corneal nerve damage and ocular surface inflammation have not been systematically evaluated. Our study aimed to investigate clinical and inflammatory changes in the ocular surface of insulin-independent type II diabetic patients in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Participants are diagnosed with dry eye according to the TFOS DEWS II diagnostic criteria: (a) OSDI questionnaire ≥13, (b) Non-invasive tear breakup time (NITBUT) <10 s, (c) ocular surface staining >5 corneal spots, greater than nine conjunctival spots (The presence of two or more criteria was used to establish a positive DE diagnosis).
* Age ≥ 18

Exclusion Criteria:

* Active ocular infection, such as infectious, viral, chlamydial, or immunologic conjunctivitis
* A history of ocular surgery that might affect the corneal or tear film, such as corneal refractive surgery, keratoplasty, cataract surgery, or ocular laser surgery
* Long-term contact lens wear
* Other ocular diseases being treated might affect the corneal or tear film: such as glaucoma, dacryocystitis, uveitis, and pterygium.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at the Department of Ophthalmology, HESH.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MMP-9 | Baseline
  MMP-9 was measured using an immunochromatography assay by collecting 1ul tear samples from the lateral canthus using a capillary tear collector. To assess the concentration of MMP-9 in the tear samples, a commercial reagent card (S05B, Seinda Biomedical Corporation, Guangdong, China) based on colloidal gold and immunochromatographic analysis was utilized. 1ul tear sample was placed in the sampling hole on the reagent card, followed by three drops of diluent in the dilution hole. The reagent card was loaded into the proprietary analyzer, and 15 minutes later, the MMP-9 concentration was measured

SECONDARY OUTCOMES:
Non-invasive tear break-up time | Baseline
  Changes in non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
Conjunctival hyperemia (RS score) | Baseline
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen
Quality of meibum grade | Baseline
  Meibum quality will be assessed under a slit-lamp: Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum).
Expressibility of meibum grade | Baseline
  Meibum expressibility will be assessed under a slit-lamp:
  Eight meibomian glands in the middle part will be evaluated on a scale of 0 to 3 (0 denoted that all glands expressible;
  1 denoted that 3 to 4 glands expressible; 2 denoted those 1 to 2 glands expressible; and 3 denoted that no glands were expressible). The overall score was computed using the mean scores of these eight glands.
Conjunctivocorneal epithelial staining grade | Baseline
  Conjunctivocorneal epithelial staining will be assessed under a slit-lamp:
  Conjunctivocorneal epithelial staining will be assess corneal and conjunctival epithelium damage. Double vital staining approach with two microliters of a preservative-free solution containing 1% lissamine green and 1% sodium fluorescein will be instilled in the conjunctival sac. The eye will be sectioned into three equal pieces (temporal conjunctiva, cornea, and nasal conjunctiva). Each region receives a maximum staining score of three points and a minimum of zero points. The combined scores from all three parts were then recorded on a scale ranging from 0 (normal) to 9 (severe)
Tear Film Lipid Layer | Baseline
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
OSDI Score | Baseline
  Chinese translated, and validated OSDI (Allergan Inc, Irvine, USA) version will beused to assess and quantify DE symptom. The 12 items of the questionnaire can be tabulated into a score that ranges from 0 (no symptoms) to 100 (severe symptoms) points
Tear meniscus height (TMH) | Baseline
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded
Corneal nerves and immune/inflammatory cells change | Baseline
  HRT III RCM, (Heidelberg Engineering GmbH, Dossenheim, Germany) will be used to record corneal nerves and immune/inflammatory cells change.
Retinal morphology | Baseline
  A scanning laser ophthalmoscope (TRC-NW300, Topcon, Tokyo, Japan) will be used to examine and record the retinal morphology, and deep learning software will be used to analyze the vascular changes of the subjects.
Central corneal sensitivity | Baseline
  Central corneal sensitivity will be measured using a Cochet-Bonnet esthesiometer (Luneau Technology Operations, France), which stimulates the cornea with a nylon monofilament. The stiffness of the filament is adjusted by altering the length (0-6cm) of the filament with a slider on the side of the pen
Corneal endothelium | Baseline
  Corneal endothelium of all patients will be photographed by contactless specular microscopy (SM) device (EM-4000; Tomey Corporation, Japan) by the same observer. The unit of cell density was evaluated as mm2
Thermal imaging: Ocular surface temperature (OST) | Baseline
  All measurements were taken in the same room with controlled temperature and humidity. Prior to ocular thermography or other tests, participants were acclimatized to the room for 20 minutes. Morgan and colleagues described the following criteria for recording OST: The patients were instructed to blink normally, close their eyes for 3 seconds, and the first image was captured soon after the eyelids opened. The temperature was taken in the central cornea, which was defined as a circular area 4 mm in diameter in the middle of the cornea

CONTACTS AND LOCATIONS:
Overall Officials: Guanghao Qin, Study Chair — He Eye Hospital
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Nentwich MM, Ulbig MW. Diabetic retinopathy - ocular complications of diabetes mellitus. World J Diabetes. 2015 Apr 15;6(3):489-99. doi: 10.4239/wjd.v6.i3.489. PMID 25897358
- [Background] Zhou Q, Yang L, Wang Q, Li Y, Wei C, Xie L. Mechanistic investigations of diabetic ocular surface diseases. Front Endocrinol (Lausanne). 2022 Dec 16;13:1079541. doi: 10.3389/fendo.2022.1079541. eCollection 2022. PMID 36589805
- [Background] Vieira-Potter VJ, Karamichos D, Lee DJ. Ocular Complications of Diabetes and Therapeutic Approaches. Biomed Res Int. 2016;2016:3801570. doi: 10.1155/2016/3801570. Epub 2016 Mar 28. PMID 27119078
- [Background] Bu Y, Shih KC, Tong L. The ocular surface and diabetes, the other 21st Century epidemic. Exp Eye Res. 2022 Jul;220:109099. doi: 10.1016/j.exer.2022.109099. Epub 2022 May 1. PMID 35508213
- [Background] Sima AA. Review: pathogenesis, progression, and therapeutic intervention of diabetic neuropathy. J Ocul Pharmacol. 1992 Summer;8(2):173-81. doi: 10.1089/jop.1992.8.173. No abstract available. PMID 1506758
- [Background] Alves Mde C, Carvalheira JB, Modulo CM, Rocha EM. Tear film and ocular surface changes in diabetes mellitus. Arq Bras Oftalmol. 2008 Nov-Dec;71(6 Suppl):96-103. doi: 10.1590/s0004-27492008000700018. PMID 19274419
- [Background] Kesarwani D, Rizvi SWA, Khan AA, Amitava AK, Vasenwala SM, Siddiqui Z. Tear film and ocular surface dysfunction in diabetes mellitus in an Indian population. Indian J Ophthalmol. 2017 Apr;65(4):301-304. doi: 10.4103/ijo.IJO_939_15. PMID 28513494
- [Background] Naik K, Magdum R, Ahuja A, Kaul S, S J, Mishra A, Patil M, Dhore DN, Alapati A. Ocular Surface Diseases in Patients With Diabetes. Cureus. 2022 Mar 22;14(3):e23401. doi: 10.7759/cureus.23401. eCollection 2022 Mar. PMID 35495002
- [Background] Bron AJ, de Paiva CS, Chauhan SK, Bonini S, Gabison EE, Jain S, Knop E, Markoulli M, Ogawa Y, Perez V, Uchino Y, Yokoi N, Zoukhri D, Sullivan DA. TFOS DEWS II pathophysiology report. Ocul Surf. 2017 Jul;15(3):438-510. doi: 10.1016/j.jtos.2017.05.011. Epub 2017 Jul 20. PMID 28736340
- [Background] Dammak A, Pastrana C, Martin-Gil A, Carpena-Torres C, Peral Cerda A, Simovart M, Alarma P, Huete-Toral F, Carracedo G. Oxidative Stress in the Anterior Ocular Diseases: Diagnostic and Treatment. Biomedicines. 2023 Jan 20;11(2):292. doi: 10.3390/biomedicines11020292. PMID 36830827
- [Background] Qin G, Chen J, Li L, Qi Y, Zhang Q, Wu Y, You Y, Yang L, Moore J, Xu L, He W, Yu S, Pazo EE, He X. Relationship between ocular surface pain and corneal nerve loss in dry eye diabetics: a cross-sectional study in Shenyang, China. BMJ Open. 2023 Sep 26;13(9):e076932. doi: 10.1136/bmjopen-2023-076932. PMID 37751961
- [Background] Bahabayi A, Yang N, Xu T, Xue Y, Ma L, Gu X, Wang Y, Jia K. Expression of Matrix Metalloproteinase-2,-7,-9 in Serum during Pregnancy in Patients with Pre-Eclampsia: A Prospective Study. Int J Environ Res Public Health. 2022 Nov 4;19(21):14500. doi: 10.3390/ijerph192114500. PMID 36361378